CLINICAL TRIAL: NCT02846870
Title: Visually Enhanced Education About Prostate Cancer (VEEP-C): A Randomized Controlled Trial
Brief Title: Visually Enhanced Education About Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Austin Kirschner, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC RAD 1646; NCI-2016-00777 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Education (Active Comparator): Patients receive standard-of-care prostate cancer radiation oncology consultation.
  Interventions: Other: Standard prostate cancer education presentation
- Visually Enhanced Education (Experimental): Patients receive a visually enhanced prostate cancer educational Powerpoint presentation including prostate anatomy, pathologic results, surgical options, radiation therapy, and prognosis with pictographs during radiation oncology consultation.
  Interventions: Other: Visually enhanced prostate cancer educational presentation

INTERVENTIONS:
Other: Visually enhanced prostate cancer educational presentation — Receive visually enhanced prostate cancer educational presentation
  Arms: Visually Enhanced Education
Other: Standard prostate cancer education presentation — Receive standard prostate cancer education presentation
  Arms: Standard Education

SUMMARY:
This randomized clinical trial studies how well visually enhanced education works in improving prostate cancer and treatment knowledge in patients with prostate cancer that has not spread to other places in the body. Visually enhanced education includes pictures, drawings, and photos, may help doctors better convey information about radiation and prostate cancer to patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Our goal is to conduct a randomized controlled trial to determine the impact of a visual presentation in the context of a radiation oncologist's discussion with patient during consultation on patient satisfaction at end of consultation visit and at end of treatment, on anxiety at start of treatment, on decision regret following treatment, and on perception of side effects following treatment. Of note, the attending radiation oncologist will be responsible for reviewing the Powerpoint presentation with the patient, taking time to answer any questions that the patient has

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM A (STANDARD EDUCATION): Patients receive a standard prostate cancer radiation oncology consultation.

ARM B (VISUAL ENHANCED EDUCATION): Patients receive a visually enhanced prostate cancer educational Powerpoint presentation including prostate anatomy, pathologic results, surgical options, radiation therapy, and prognosis with pictographs during radiation oncology consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have non-metastatic, biopsy proven prostate cancer
* Must be referred to radiation oncology clinic

Exclusion Criteria:

* Prior surgery or radiation therapy for prostate cancer
* Patients who are blind are excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Decision-Regret - based on Ottawa scale | Up to 12 weeks
  Sample size was determined based on this primary outcome - with estimated mean of 16 in Arm A and mean of 8 in Arm B, with standard deviation of 15, with 80% power and alpha of 0.05.

SECONDARY OUTCOMES:
Satisfaction - SCA | baseline, end of treatment, and long-term follow-up
Symptoms based on EPIC-26 short form | baseline, end of treatment, and long-term follow-up
Anxiety - Memorial MAX-PC scale | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Austin Kirschner, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT02846870/ICF_000.pdf